CLINICAL TRIAL: NCT04009616
Title: Effect of Aloe Vera Mouthwashes on Plaque and Gingivitis Indices in Children (Clinical Randomized Controlled Trial)
Brief Title: Effect of Aloe Vera Mouthwashes on the Oral Health of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UDDS-Pedo-01-2020
Record Dates: First submitted 2019-06-25; First posted 2019-07-05 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Oral Health
Keywords: Aloe vera mouthwash

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aloe Vera mouthwash (Experimental): plaque accumulation and gingivitis will be evaluated before and after giving aloe vera mouthwash by studying plaque, gingival and bleeding indices.
  the plaque will be accumulated for 3 days "accumulation phase" before applying aloe vera mouthwash for 5 days "rinsing phase".
  Interventions: Drug: Aloe Vera mouthwash
- Chlorhexidine mouthwash (Experimental): plaque accumulation and gingivitis will be evaluated before and after giving chlorhexidine mouthwash by studying plaque, gingival and bleeding indices.
  the plaque will be accumulated for 3 days "accumulation phase" before applying chlorhexidine mouthwash for 5 days "rinsing phase".
  Interventions: Drug: Chlorhexidine mouthwash
- Placebo mouthwash (Placebo Comparator): plaque accumulation and gingivitis will be evaluated before and after giving placebo mouthwash by studying plaque, gingival and bleeding indices.
  the plaque will be accumulated for 3 days "accumulation phase" before applying placebo mouthwash for 5 days "rinsing phase".
  Interventions: Drug: Placebo mouthwash

INTERVENTIONS:
Drug: Aloe Vera mouthwash — rinsing with aloe vera mouthwash for 5 days.
  Arms: Aloe Vera mouthwash
Drug: Chlorhexidine mouthwash — rinsing with chlorhexidine mouthwash for 5 days.
  Arms: Chlorhexidine mouthwash
Drug: Placebo mouthwash — rinsing with placebo mouthwash for 5 days.
  Arms: Placebo mouthwash

SUMMARY:
Prevention of dental problems by controlling plaque is the best solution to maintain oral health and prevent high cost of dental treatments. Home oral care is the cornerstone in removing plaque and therefore controlling tooth decay and gum disease. Unfortunately, complete plaque removal is difficult to achieve by mechanical methods alone.

For effective plaque control antiplaque agents such as chlorhexidine mouthwash is necessary. Chlorhexidine has shown distinct advantage, but it has many side effects such as staining of the teeth and the tongue, altered taste sensation, and increased calculus formation often deters its use for long periods.

Recently the use of herbal mouthwashes is rising due to the widespread awareness that natural substances have less side effects and lower economic cost. Of various plant extracts used as a base for mouthwashes, aloe vera deserves a special attention as it has recently been introduced in dentistry after years of use in medicine field.

Many recent studies stated that aloe vera mouthwashes has shown efficiency in plaque control and prevention of gingivitis, but there is a need for more studies to determine the best protocols regarding concentration and frequency of its use. A review of the literature shows that there is no randomized controlled trials evaluating its efficiency in plaque control and prevention of gingivitis in children, which is the main purpose of this study.

DETAILED DESCRIPTION:
The crossover design will be adopted in this study, i.e. the three types of mouthwashes (experimental "aloe Vera", positive control "chlorhexidine", negative control "placebo") will be utilized for all participants, with an equal (5) days application period for each type of mouthwashes and a wash-out period of (12) days between each type to ensure the elimination of the effects of a mouthwash before moving to the next one.

The evaluation areas selected for the study comprised the central maxillary incisors and the first maxillary molars.

A special plaque guard will be fabricated to cover the evaluated teeth and their gingival margins, this plaque guard will prevent plaque removal of the evaluated teeth and facilitate localized plaque accumulation and the resultant gingivitis if any.

At the start of the study, all participants will be instructed on how to brush their teeth properly and continue their regular oral hygiene.

All subjects will be instructed to wear the plaque guards every time they cleaned their teeth, so that they will not brush the maxillary incisors and the maxillary first molars. This phase "the accumulation phase" will last for 3 days, and then the subjects will be recalled to assess the difference in plaque accumulation on the 5th day.

The following indices will be studied: Plaque index (PI) to assess the plaque accumulation, gingival index (MGI),and bleeding index (BI)to assess gingivitis. These indices will be recorded at the first and in the 3th day. The "rinsing phase" will begin from the morning of day 4 and last for 5 days.

15 ml of rinsing solution will be given to each subject who is not aware of what type of mouthwash he/she is receiving. Along with each bottle of mouthwash, a 10 ml syringe will be used to facilitate determining correct dosage. The subjects will be asked to rinse with 15 ml of the solution for 1 min, once daily. Intake of food and/or drinks will not be allowed for 2 hours after rinsing. The subjects will be recalled for evaluation of plaque accumulation once the "rinsing phase" is completed on 8th day.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ages between (8 - 12) years.
2. Healthy children without any systemic medical conditions.
3. Good oral health (no manifestations of oral diseases on the mucous membranes).
4. The presence of the maxillary first permanent molars and the maxillary central incisors.
5. No caries on the buccal and lingual surfaces of the teeth.
6. Cooperative children (positive or definitely positive on Frankl's behavior rating scale).
7. The patient has the physiological ability to use the mouthwashes, This will be confirmed by asking the child's parent first and then test his/her ability to rinse with water before being enrolled in the study.

Exclusion Criteria:

1. Children with systemic medical conditions.
2. Patients undergoing current dental or orthodontic treatment.
3. Patients who used any other mouthwash during the study period or were given antibiotic therapy within 2 weeks before starting the study or corticosteroids within 30 days before starting the study.
4. Patients who use removable prosthetic or orthodontic appliances.
5. Patients who have gingival pockets more than (3) mm or advanced gingival diseases.
6. Fluorescent patients.
7. Patients who have a sensitivity story for any element of the mouthwashes used in the study.
8. Patients who underwent an extraction within two weeks of starting the study.
9. Patient lack of commitment toward follow-up appointments.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Effect of Aloe vera mouthwashes on plaque index | before accumulation phase (at the 1st day), before rinsing phase (at the 3rd day) and after rinsing phase (at the 8th day)
  this variable will be measured by calculating the difference between the index studied at the beginning and end of the experimental phase, to evaluate children's oral health and know the probability to have caries later.
Effect of Aloe vera mouthwashes on gingival index | before accumulation phase (at the 1st day), before rinsing phase (at the 3rd day) and after rinsing phase (at the 8th day)
  this variable will be measured by calculating the difference between the index studied at the beginning and end of the experimental phase, to evaluate children's gingival health and know the probability to have gingivitis later.
Effect of Aloe vera mouthwashes on gingival bleeding index | before accumulation phase (at the 1st day), before rinsing phase (at the 3rd day) and after rinsing phase (at the 8th day)
  this variable will be measured by calculating the difference between the index studied at the beginning and end of the experimental phase, to evaluate children's gingival health and know the probability to have gingivitis later.

SECONDARY OUTCOMES:
the level of receptivity and discomfort and side effects of the Aloe vera mouthwashes. | at the end of each mouthwash experimental phase (8th day)
  Assessment will be performed using questionnaire that includes Visual Analog Scale (VAS) for each question, the scale has a minimum scale of 0 (no discomfort) and a maximum scale of 100 (maximum discomfort).

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Adnan Alnouri, DDS, Msc Student, Principal Investigator — Department of Pediatric Dentistry, Faculty of Dental Medicine, Damascus University, Damascus, Syria; Chaza Kouchaji, Professor, Study Chair — Department of Pediatric Dentistry, Faculty of Dental Medicine, Damascus University, Damascus, Syria; Abdul Hakim Nattouf, Professor, Study Chair — Department of Pharmaceutics and Pharmaceutical Technology, Faculty of Pharmacy, Damascus University, Damascus, Syria
Locations (1):
- Faculty of Dental Medicine, Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ajmera N, Chatterjee A, Goyal V. Aloe vera: It's effect on gingivitis. J Indian Soc Periodontol. 2013 Jul;17(4):435-8. doi: 10.4103/0972-124X.118312. PMID 24174720
- [Background] Gupta RK, Gupta D, Bhaskar DJ, Yadav A, Obaid K, Mishra S. Preliminary antiplaque efficacy of aloe vera mouthwash on 4 day plaque re-growth model: randomized control trial. Ethiop J Health Sci. 2014 Apr;24(2):139-44. doi: 10.4314/ejhs.v24i2.6. PMID 24795515
- [Background] Manipal S, Hussain S, Wadgave U, Duraiswamy P, Ravi K. The Mouthwash War - Chlorhexidine vs. Herbal Mouth Rinses: A Meta-Analysis. J Clin Diagn Res. 2016 May;10(5):ZC81-3. doi: 10.7860/JCDR/2016/16578.7815. Epub 2016 May 1. PMID 27437366
- [Background] Pilloni A, Pizzo G, Barlattani A, Di Lenarda R, Giannoni M, Guida L, Levrini L, Majorana A, Polimeni A. Perceived and measurable performance of daily brushing and rinsing with an essential oil mouthrinse. Ann Stomatol (Roma). 2010 Jul;1(3-4):29-32. Epub 2011 Feb 13. PMID 22238712
- [Background] Saha S, Mohammad S, Saha S, Samadi F. Efficiency of traditional chewing stick (miswak) as an oral hygiene aid among Muslim school children in Lucknow: A cross-sectional study. J Oral Biol Craniofac Res. 2012 Sep-Dec;2(3):176-80. doi: 10.1016/j.jobcr.2012.10.009. Epub 2012 Oct 24. PMID 25737862